CLINICAL TRIAL: NCT01647633
Title: Effects of AkPharma's Calcium Glycerophosphate Nasal Spray Wash on Patient-Perceived Breathing Comfort
Brief Title: Effects of AkPharma's Calcium Glycerophosphate Nasal Spray Wash
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: AkPharma Inc. (Industry)
Responsible Party: Principal Investigator, Edward Schulman, MD, PI, Drexel University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AkP 010112A
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Allergic Rhinitis
Keywords: rhinitis; stuffy nose; congestion; Sneezing
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis; Nasal Obstruction; Sneezing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Calcium Glycerophosphate Nasal Wash (Experimental): Nasal spray wash twice daily and up to four additional times per day as needed for nasal allergy symptoms
  Interventions: Other: Calcium Glycerophosphate Nasal Spray Wash

INTERVENTIONS:
Other: Calcium Glycerophosphate Nasal Spray Wash — Nasal wash two to six times per day

SUMMARY:
Over 20 million Americans have allergic nasal symptoms including stuffiness, sneezing and a "runny" nose. AkPharma's Calcium Glycerophosphate used as a nasal spray wash is believed to improve these symptoms without side effects common to over the counter and prescription medication. It is hypothesized that Calcium Glycerophosphate will have a perceived improvement in breathing comfort.

DETAILED DESCRIPTION:
Subjects will be screened for inclusion and exclusion criteria and consented if they fit the same criteria. They will be instructed on keeping a nasal diary of symptoms "runny, itchy, congestion, sneezing, voice changes and throat clearing". They will have blood drawn for allergy testing. After a 1 week run-in, subjects will return their diary. If they still qualify based on the diary they will have baseline labs drawn and baseline breathing test (Spirometry) performed. They will also have a nasal wash and specimen collection performed. They will be instructed on use of the nasal wash. There will be three more weekly visits before study conclusion which will include diary submission, Spirometry and nasal wash and specimen collection. On the final visit blood will again be collected as well.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female 18-80 years of age
* Twelve months or more of allergic rhinitis symptoms
* Allergic antibodies to perennial aeroallergens to be confirmed by blood draw

Exclusion Criteria:

* Intranasal or systemic glucocorticosteroids within one month of study entry
* Intranasal cromolyn for 2 weeks prior to study
* Intranasal or systemic antihistamine for 3 days prior to the study
* Loratadine for ten days prior to study
* History of rhinitis medicamentosa
* Planned travel outside the study area that will inhibit study follow-up visits

  _Persons with Asthma with more than 2 episodes per week or month of nighttime awakenings
* Persons with Known sensitivity to Calcium or phosphorus supplements
* Persons taking antihistamine treatment intermittently. (Chronic steady use throughout study is acceptable)
* Immunomodulatory or cytotoxic drugs
* Clinically significant uncontrolled disease that in the opinion of the investigator would put the subject at risk or may confound the study interpretation
* Persons with hypercalcemia
* Persons whose nasal obstruction(s) would be significant to obstruct air flow
* Persons who are employees of Investigator or AkPharma or whose spouse, parent, child or sibling is employee of investigator
* Pregnant persons or persons planning to conceive/inseminate partner during study or for one month after

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-05; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Nasal Symptom Diary | 28 days
  Perceived improved comfort breathing is anticipated as primary outcome

SECONDARY OUTCOMES:
Spirometry | 21 days
  Anticipate change in spirometry

CONTACTS AND LOCATIONS:
Overall Officials: Edward S Schulman, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine, Philadelphia, Pennsylvania, United States